CLINICAL TRIAL: NCT04895527
Title: Air-test as a Predictor of Pulmonary and Systemic Complications After Laparoscopic Surgery
Status: Completed | Type: Observational
Sponsor: Dr. Negrin University Hospital (Other)
Responsible Party: Principal Investigator, Ángel Becerra, Principal Investigator, Dr. Negrin University Hospital
Other Study IDs: Airtest-Negrín
Record Dates: First submitted 2021-05-17; First posted 2021-05-20 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Postoperative Complications
Keywords: airtest; atelectasis; postoperative period; complications
MeSH Terms: conditions — Postoperative Complications; Pulmonary Atelectasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
One of the main risk factors for the development of postoperative pulmonary complications (PPC) in postsurgical patients is the persistence of atelectasis during this period. Therefore, it would be of great clinical interest to establish a causal relationship between postoperative atelectasis and the development of PPC, as well as having a relatively precise, simple and non-invasive method to rapidly diagnose these atelectasis.

A prospective observational study will be carried out including all patients undergoing scheduled laparoscopic surgery, excluding pregnant women or women in the period of lactation, patients with moderate - severe acute respiratory distress syndrome, heart failure, need for mechanical ventilation during the 15 days prior to surgery or with a history of cardiothoracic surgery. Demographic variables (age, sex, weight, BMI), preoperative data (presence of allergies, cardiovascular risk factors, personal cardiopulmonary history, presence of toxic habits, baseline peripheral oxygen saturation, ASA classification, ARISCAT and frailty markers will be collected - Fried phenotype, scale clinical frailty and FRAIL scale -) and intraoperative (duration of the procedure, recruitment maneuvers). At 30 postoperative days the history will be reviewed clinic of the patients and the postoperative complications will be collected. Main objective: to demonstrate the veracity of the air-test in the prevention of pulmonary or other systemic complications in patients undergoing laparoscopic surgery.

Secondary objectives:

* Measure the incidence of positive results in the air-test.
* Demonstrate the correlation between the performance of recruitment maneuvers and a negative score in the air-test
* Demonstrate the correlation between the degree of frailty of the patients and a positive score in the air-test.

DETAILED DESCRIPTION:
The persistence of postsurgical atelectasis is potentially associated with complications such as pneumonia, acute respiratory distress, and hypoxemia. This promotes other systemic complications such as myocardial ischemia or healing defects, negatively affecting morbidity, healthcare costs, and postoperative survival. Pre and intraoperative hemoglobin saturation levels are an independent risk factor for postoperative pulmonary complications. The airtest, based on the measurement of peripheral oxygen saturation (SpO2) with ambient air in the early postoperative period, is a useful tool in the prevention of moderate-severe pulmonary postsurgical complications.

One of the main risk factors for the development of postoperative pulmonary complications (PPC) in postsurgical patients is the persistence of atelectasis during this period. Therefore, it would be of great clinical interest to establish a causal relationship between postoperative atelectasis and the development of PPC, as well as having a relatively precise, simple and non-invasive method to rapidly diagnose these atelectasis.

A prospective observational study will be carried out including all patients undergoing scheduled laparoscopic surgery, excluding pregnant women or women in the period of lactation, patients with moderate - severe acute respiratory distress syndrome, heart failure, need for mechanical ventilation during the 15 days prior to surgery or with a history of cardiothoracic surgery. Demographic variables (age, sex, weight, BMI), preoperative data (presence of allergies, cardiovascular risk factors, personal cardiopulmonary history, presence of toxic habits, baseline peripheral oxygen saturation, ASA classification, ARISCAT and frailty markers will be collected - Fried phenotype, scale clinical frailty and FRAIL scale -) and intraoperative (duration of the procedure, parameters, recruitment maneuvers). At 30 postoperative days the history will be reviewed clinic of the patients and the postoperative complications will be collected. Main objective: to demonstrate the veracity of the air-test in the prevention of pulmonary or other systemic complications in patients undergoing laparoscopic surgery at the Doctor Negrín University Hospital of Gran Canaria.

Secondary objectives:

* Measure the incidence of positive results in the air-test.
* Demonstrate the correlation between the performance of recruitment maneuvers and a negative score in the air-test
* Demonstrate the correlation between the degree of frailty of the patients and a positive score in the air-test.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing scheduled laparoscopic surgery

Exclusion Criteria:

* Pregnant or lactating women.
* Presence of moderate to severe acute respiratory distress.
* Patients suffering from heart failure.
* Patients undergoing invasive mechanical ventilation during the 15 days prior to surgery.
* Patients with a history of cardiothoracic surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing scheduled laparoscopic surgery will be included and informed consent will be asked to perform air-test postoperatively.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Postoperative pulmonary complications | 30 days postoperatively
  to demonstrate the veracity of the air-test in the prevention of pulmonary complications in patients undergoing scheduled laparoscopic surgery
Postoperative systemic complications | 30 days postoperatively
  to demonstrate the veracity of the air-test in the prevention of systemic complications in patients undergoing scheduled laparoscopic surgery

SECONDARY OUTCOMES:
Incidence of positive air-test | 4 hours postoperatively
  to detect the prevalence of patients showing positive in the air-test in the postoperative period after scheduled laparoscopic surgery
Recruitment maneuvers and air-test | from the intraoperative period (recruitment maneuvers) until 4 hours postoperatively
  to demonstrate the correlation between the performance of recruitment maneuvers and a negative score in the air-test

CONTACTS AND LOCATIONS:
Overall Officials: Ángel Ángel, MD, Principal Investigator — Hospital Universitario de Gran Canaria Doctor Negrín
Locations (1):
- Ángel Becerra, Las Palmas de Gran Canaria, Las Palmas, Spain

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data can be available after request to the principal investigator